CLINICAL TRIAL: NCT00879632
Title: Brain Derived Neurotrophic Factor as a Predictor of Response to Treatment in Bipolar Depression and Mania: 16-weeks Follow-up Study
Brief Title: Brain Derived Neurotrophic Factor as a Predictor of Response to Treatment in Bipolar Depression and Mania
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Flavio Kapczinski, Hospital de clinicas de porto alegre
Other Study IDs: 07456
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: BIPOLAR DISORDER
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SERUM, DNA, PLASMA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: TREATMENT AS USUAL
- 2: CONTROLS

SUMMARY:
There is sound evidence that quetiapine is effective in the treatment of manic and depressive episodes associated with Bipolar Disorder (BD) (Yatham et al 2006). However, even with the development of effective new treatment options, not all patients respond to treatments available. Biological markers have been investigated as predictors of response to treatment and of remission of symptoms. This would explain in part the individual's differences in the response to treatment, taking into account the genetic variability plus environmental factors influencing specific biological markers. A potential biological marker of response to treatment in BD would be the levels of neurotrophins, as they are, in fact, altered during acute mood episodes (Cunha et al 2006). Among neurotrophins, the Brain-Derived Neurotrophic Factor (BDNF) has been repeatedly and consistently reported to be associated with BD physiopathology (Post 2007). Furthermore, medications that are known to be effective in BD, like lithium and divalproex, increase BDNF levels.

DETAILED DESCRIPTION:
There is sound evidence that quetiapine is effective in the treatment of manic and depressive episodes associated with Bipolar Disorder (BD) (Yatham et al 2006). However, even with the development of effective new treatment options, not all patients respond to treatments available. Biological markers have been investigated as predictors of response to treatment and of remission of symptoms. This would explain in part the individual's differences in the response to treatment, taking into account the genetic variability plus environmental factors influencing specific biological markers. A potential biological marker of response to treatment in BD would be the levels of neurotrophins, as they are, in fact, altered during acute mood episodes (Cunha et al 2006). Among neurotrophins, the Brain-Derived Neurotrophic Factor (BDNF) has been repeatedly and consistently reported to be associated with BD physiopathology (Post 2007). Furthermore, medications that are known to be effective in BD, like lithium and divalproex, increase BDNF levels. Diverse sources of evidence provide support to the alteration of BDNF in mood disorders:

* Patients with major depressive disorder showed lower levels of BDNF and the treatment with antidepressants recovered those levels back to normal. (Gonul et al 2005).
* Studies with brain tissue (post-mortem) showed that BDNF levels were decreased only on those who were not on antidepressants. (Karege et al 2002).
* The polymorphism of BDNF gene was associated with response to treatment with lithium during maintenance phase. (Rybakowski et al. 2005).
* Our group showed that BDNF levels are decreased during mania and depression, but not during remission (Cunha et al 2006, Machado-Vieira et al. 2007). Therefore, BDNF appear to be involved in the mechanisms of acute mood episodes.
* Treatment with mood stabilizers, such as lithium and divalproex, increase BDNF levels (Frey et al. 2006).

Prediction of drug treatment response based on variation in genetic make up is a rapidly growing area. However, few studies examined the association between single nucleotide polymorphisms and drug response in bipolar disorder. The design of this study offers a unique opportunity to examine genetic predictors of drug response. Interestingly, a single nucleotide polymorphism at nucleotide196 (G/A) in the human BDNF gene at codon 66 (Val66Met) have been reported to be associated with a predisposition to BD in family-based studies (Rybakowski et al 2006, Green et al 2006). In humans, this polymorphism produces a valine - to - methionine substitution in the proBDNF protein and reduces the trafficking and secretion of BDNF protein. This is relevant because it has been estimated that 20-30% of the human population is heterozygous for the Met polymorphism of BDNF. Furthermore, there are consistent findings in BD regarding the association of Val66Met polymorphism of BDNF gene with prefrontal cognitive impairment, which was recently confirmed in a large sample of bipolar subjects (Rybakowski et al 2006). In addition, crosssectional studies showed that the polymorphism of BDNF gene (Val66Met) was associated with response to lithium prophylaxis, but findings were not universal (Rybakowski et al 2005, Masui et al 2006). However, there is a need for prospective studies in order to confirm these findings. It is possible that a single polymorphism of BDNF gene would have a negative impact of BDNF levels and, consequently, a negative impact in the response to treatment.

Despite consistent evidence of changes in BDNF levels during mood episodes and treatment, one important aspect remains unknown: Whether the change in BDNF levels is required for treatment response and whether the magnitude of change happens in portion with the response to treatment and remission of symptoms.

The hypothesis for this project is that those patients who have a good response to treatment are the same ones who show the greater increase in BDNF levels earlier in the course of treatment, and who are less likely to present a polymorphism of BDNF gene. Given this context, we aim to investigate BDNF levels prospectively in patients with BD, before, during and after the treatment with quetiapine and compare measures with response to treatment, as indicated by remission in symptoms. We also aim to investigate the polymorphism of BDNF gene (Val66Met) and its correlation with BDNF serum levels and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. A diagnosis of Bipolar Disorder I by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition revised (DSM-IV-TR)
3. Males and females aged 18 to 65 years
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotrophin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study
6. Currently experiencing a manic, depressive or mixed mood episode, according to DSM-IV-TR. Patients must have a clear DSM-IV diagnosis, confirmed by SCID interview (Structured Clinical Interview for DSM disorders).

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
5. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
6. Currently on psychotropic medication or administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation. Wash-out of minimum of 2 weeks will be required for intake. Fluoxetine use or depot antipsychotics will require 6 weeks of wash-out prior to intake.
7. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
8. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
9. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
10. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
11. Involvement in the planning and conduct of the study
12. Previous enrolment in the present study.
13. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
14. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bipolar disorders patients during acute mania or depression using treatment as usual
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton depression raing scale and young mania rating scale | 16 weeks

SECONDARY OUTCOMES:
Serum BDNF levels as predictor of response to treatment | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: FLAVIO KAPCZINSKI, MD, PHD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil